CLINICAL TRIAL: NCT06695325
Title: Comparability of Analyte Levels, Patient Acceptance and Health Economics Between Self-collected Capillary Blood (In-clinic and Home) and Professionally Collected Venous Blood for HbA1c, Lipids and Thyroid Function in Diabetic Patients
Brief Title: Convenient Home Access for Routine Monitoring in Diabetes (Charm-D Study)
Acronym: CHARM-D
Status: Recruiting | Type: Observational
Sponsor: Tameside General Hospital (Other)
Collaborators: Roche Diagnostic Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: Tameside003; Roche (Other Grant/Funding Number: Roche)
Record Dates: First submitted 2024-11-14; First posted 2024-11-19 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Diabetes Mellitus
Keywords: Home monitoring; HbA1c; Thyroid function; Lipids
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with type 1 and type 2 diabetes will be invited to take part in this study: Patients will be asked to have a HbA1c test in the clinic with a venous draw and then either fingerprick or upper arm draw. They will do the latter again at home.
  Interventions: Diagnostic Test: HbA1c test

INTERVENTIONS:
Diagnostic Test: HbA1c test — Patients will be asked to have a HbA1c test in the clinic with a venous draw and then either fingerprick or upper arm draw. They will do the latter again at home.

SUMMARY:
Diabetes mellitus is a global problem and regular monitoring of blood sugar control is important to reduce the risk of complications secondary to poor sugar control. To assess control a simple blood test is undertaken called the HbA1c. This test gives an assessment of the person's sugar control over the previous 3 months and needs to be done regularly so that changes can be made to their treatment. The HbA1c test is routinely performed in clinic and blood taken from a vein in the arm using a needle and syringe. This involves travelling to the clinic, taking time off work and expense to the patient. Many times and for the above reasons patients do not attend the clinic and therefore do not have the HbA1c performed. Therefore the clinician will not know how their diabetes is doing and also they will not be able to make changes to the patient's diabetes treatment.

In this study we would like to assess home monitoring of diabetes by doing the HbA1c at home and sent to the laboratory. At the same time we will be checking the patient's blood cholesterol (lipids) levels and thyroid function (to assess if the thyroid gland which is in the neck, is making adequate hormones).

In the study the patient will first visit the clinic where blood will be taken from the arm as is done in routine clinical care. Then the patient will take blood himself/herself either from the finger (finger prick as is done when a patient checks their own blood glucose) or from the upper arm using a device that will be applied to the skin and blood will be collected in a small tube attached to the device. Half the patients will be asked to do a finger prick test and the other half will do the upper arm skin blood draw. The patient will be asked to fill a questionnaire, this is to understand their experience with the blood self-collection and how they classify it in comparison with the routine clinical care.

The patient will then go home with the similar device that they used in the clinic and will be asked to do the same blood draw at home as they did in the clinic (either finger prick or upper arm blood draw). They will need to do this within 2 days of the visit to the clinic. They will then post the sample to the central laboratory in the envelope provided.

At the same time the patient will be asked to fill out a questionnaire. This is to understand the ease or difficulty of the testing at home but will also help us analyse the cost effectiveness of doing the home blood collection.

DETAILED DESCRIPTION:
BACKGROUND Diabetes management heavily relies on the regular monitoring of HbA1c levels, which provides a comprehensive picture of blood sugar control over the past two to three months. The current standard involves venous blood draws, which are performed by healthcare professionals in clinical settings. However, this method has limitations, including long waiting times and irregular check-ups due to a shortage of qualified staff. This issue is more pronounced in rural areas where access to healthcare services is limited.

Recent advancements in capillary blood collection techniques have shown that capillary blood sampling can be as accurate as venous blood sampling for certain parameters such as HbA1c, lipids, and thyroid. These findings suggest that home-based self-collection could be a viable alternative to traditional methods, offering greater convenience and accessibility for patients.

RATIONALE

The primary aim of this study is to evaluate the accuracy and feasibility of home-based self-collected capillary blood sampling in comparison to the standard venous blood collection performed by healthcare professionals. Specifically, the study will assess the accuracy accuracy of blood drawn in clinic for HbA1c levels, the lipid (cholesterol, HDL, LDL), and thyroid (TSH, fT3, fT4) compared to blod collected through self-sampling at home. Additionally, this study will evaluate patient acceptance and the economic impact of this approach.

Regular monitoring of HbA1c is crucial for diabetes management, but current venous blood draw methods often lead to long waiting times and irregular check-ups due to staff shortages. This issue is particularly pressing in rural areas with limited healthcare access. Home-based self-collection could alleviate these challenges by freeing up healthcare staff, reducing waiting times, enabling more frequent monitoring.

This study addresses a crucial gap in the current diabetes management paradigm by exploring a more convenient and accessible method for blood sample collection. By generating evidence on the method accuracy, patient acceptance, and economic impact of home-based self-collection, this research has the potential to significantly improve healthcare delivery. It can also enhance patient outcomes, particularly for those in underserved areas.

RESEARCH QUESTION/AIM(S) To compare the method accuracy for blood monitoring, the patient acceptance and consideration of health economics between self-collected capillary blood and professionally collected venous blood for HbA1c, LDL, HDL, cholesterol, TSH, fT3, and fT4.

Outcomes: see below

STUDY DESIGN Single site (tameside general hospital, Ashton under Lyne), randomised controlled trial consisting of three blood samples per patient and two questionnaires. After consent a venous blood sample will be taken by nurse in the clinic. Participants will then be randomised toperform a capillary self-collection with either an upper arm device or a finger prick device at the clinic. The capillary draw will be a self-collection, training will be provided to the participant. Participants will be asked to collect a further capillary sample outside the clinic (preferably at home), within 24 hours of the hospital appointment. Participants will be provided with a prepaid and addressed shipping package to post the sample to the laboratory. The participant will be asked to complete a short questionnaire following taking the in-clinic capillary sample as well as the outside the clinic capillary sample to provide details of the ease of use and opinions of the self-collection device compared with the standard care.

The study staff will be asked to complete a case report form to provide details on the blood collection in the clinic.

Shipping packages contain a temperature-monitoring label to enable the study team to track the sample temperature whilst in transit to the laboratory. The research nurse will activate the temperature-monitoring label in the clinic before providing the packaging to the participant. If the laboratory does not receive an outside the clinic sample within the week of collection, the research team will try to contact the participant by phone to see if there were any issues for collecting the sample. The study will assess for non-compliance/lost packages/collection failures as this will provide evidence for the usability of the 'outside the clinic' collected capillary samples. If the missing sample is due to the participant having issues with the device or sample collection, they will be invited back to the clinic for a further research visit and the sample collection process will start again, as all three samples (in clinic venous, in clinic capillary and outside the clinic capillary) are required to be analyzed at the same time for accuracy. This will be documented as a second visit with the reason for the missing sample documented. The participant will be informed about the potential for a second visit in the participant information sheet, and notified that this is optional. The research team will make three telephone attempts to contact the participant, after which, it will be noted as a collection failure.

Due to the possible low sample volume obtained by the capillary self-collection the analytes to be measured are prioritized. The focus of the study is HbA1c, followed by lipids. If sufficient sample volume is available the thyroid panel will be measured in a second measurement, however this is considered to be more exploratory.

The study aims to assess the potential health economic (HE) advantages of outside the clinic blood self-collection compared to traditional venous blood draws conducted in hospitals or general practitioners' (GP) offices.

Healthcare professionals performing blood draws in clinical settings incur costs that can be avoided if patients collect samples themselves. Additionally, patients incur expenses related to travelling to and from their GP's office or hospital, as well as potential income loss from taking time off work for healthcare visits, all of which can affect their overall health expenditures.

Samples will be posted to the laboratory INUVI located in England for processing and analysis. The laboratory will know which samples are collected with which device, as the collection tubes will be different.

Inclusion and exclusion criteria: see below

Patients A sample size of N=150 per capillary blood draw per device (total 300) was chosen to be able to show an acceptable accuracy, defined as 95% of all differences within the acceptance region and with the lower limit of the 95% CI ≥ 90%, for each analyte with at least 80% power. Sample size estimation is based on the exact binomial test.

Recruitment: From diabetes clinics at Tameside hospital. Participants will be offered £50 for participating in the study, which is to cover travel expenses for the additional research visit and a small inconvenience payment.

PI will take Informed consent from participants prior to any study procedures taking place and will provide a participant information sheet (PIS) and an overview of the study to consider participation.

Participants will be trained to use the self blood collection device, to use outside the clinic. This will be provided by the research nurses in the clinic.

Questionnaire Objectives of the study will be assessed using answers taken from the questionnaire.

1. How does the preference of patients compare for outside the clinic collection vs the standard of care?
2. Did the participant experience any side effects? how convenient was the venepuncture?.
3. How painless the self-collection was for the participant. All three questions have answers ranging from 1 to 10. All costs linked to sample collection of blood self-collection outside the clinic will be compared to the costs linked to the standard of care (venepuncture).

ETHICAL AND REGULATORY CONSIDERATIONS The CI, Professor Edward Jude, will submit an application for Research Ethics Committee. The sponsor will ensure that all relevant approvals have been granted before any trial activities commence.

To compensate, participants will be offered £50 for participating in the study, to cover travel expenses (£30) and inconvenience payment (£20).

The devices being used are CE marked and being used within their intended purpose. Devices are being provided by Roche Diagnostics International Ltd. The laboratory being used in the study has UKAS accreditation.

Due to the analytical study design no diagnosis will be made, no treatment will be initiated and no medical decision will be taken solely based on the results measured from the sample specimen. In case of out-of-normal results of the professionally collected venous sample the study team will review the results and, if appropriate, forward results to the participant's treating physician for a follow-up.

An annual progress report will not be required in accordance with the updated process, as the study is expected to run for less than two years and is recruiting in England only. On conclusion of the study, an end of study notification and final report will be submitted to the REC that provided the favourable opinion for the study. The end of study notification will be within 90 days of the study ending.

Within one year after the end of the study, the Chief Investigator will submit a final report to the REC, with the results and any publications. The end of study will be the date of the last data collection for the last participant.

Data protection and patient confidentiality Data collected during the study will kept strictly confidential and handled in accordance with the GDPR and Data Protection Act (2018). The study will obtain informed consent from the participant prior to accessing the patient's medical records. Participants will be identified by a unique study ID number once they have consented to the study. All personal identifiable information will be retained on a separate password protected database which will be stored on the secure hospital network with restricted access to the investigator and research team only. A separate linked password protected database containing the study data will be stored in a separate location on the secure hospital network system, with access restricted to the Investigator and research team only and kept securely. We will keep identifiable information for a maximum of 3 years after the study has finished. This excludes any research documents with personal information, such as consent forms, which will be archived securely at the end of the study, in accordance with the sponsors archiving requirements, before being confidentially destroyed. The sponsor's current archiving duration for this trial type is a minimum of 15 years from the end of study date. The sponsor will be the data custodian.

All data will be anonymized before being provided to Roche Diagnostics International Ltd. for analysis. No personal identifiable information will be included as part of the study results or publications.

Indemnity: The study sponsor is Tameside and Glossop Integrated care NHS Foundation Trust and NHS indemnity scheme will apply. The design of the study will be jointly indemnified by the sponsor and Roche Diagnostics International Ltd. The device will be indemnified by the manufacturer.

ELIGIBILITY:
Inclusion Criteria:

* Adult subjects aged 18 years and over at the time of signing the informed consent
* Ability to provide Informed consent
* Type I and II diabetic patient
* Ability to understand written and spoken English
* Ability to perform a blood draw at home

Exclusion Criteria:

* Aged less than 18 years of age
* Unable to provide informed consent
* Unable to perform a blood draw at home

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants will be identified and approached during a routine diabetes clinic service run by Tameside and Glossop Integrated Care NHS Foundation Trust, based at Ashton Primary Care. This is a single site study. Consent, randomisation and a venous and a capillary self-collected sample will be collected at Tameside and Glossop Integrated Care NHS Foundation Trust. A second capillary sample will be self-collected by the participant in an outside the clinic setting and posted to the central laboratory. Participants will complete a questionnaire in the clinic as well as outside the clinic. The outside the clinic questionnaire will be posted back to the research team at Tameside General Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2025-11-04 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
HbA1c | 12 months
  to evaluate the accuracy and compare HbA1c measurement in-clinic testing by venous draw by health professionals vs home-based self-collected capillary blood sampling

SECONDARY OUTCOMES:
Lipids | 12 months
  to evaluate the accuracy and compare lipid measurement in-clinic testing by venous draw by health professionals vs home-based self-collected capillary blood sampling
Thyroid function | 12 months
  to evaluate the accuracy and compare thyroid function measurement in-clinic testing by venous draw by health professionals vs home-based self-collected capillary blood sampling
Participant acceptance | 12 months
  Participant acceptability of collecting a outside the clinic capillary sample. Patients will be asked to answer questions on pain experience from venous draw vs home collection of blood sample, convenience of attending clinic for venous drwa vs home- collection and will be scored from 1-10 (Visual analo scale).
Health economics | 12 months
  Health economic value of collecting outside the clinic capillary sample versus standard of care venous draw

CONTACTS AND LOCATIONS:
Overall Officials: Edward Jude, MD FRCP, Principal Investigator — Tameside and Glossop Integrated Care NHS Foundation Trust
Locations (1):
- Tameside and Glossop Integrated Care NHS Foundation Trust, Ashton-under-Lyne, Lancs, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
All data will be kept confidential and at the study site. No patient identifiable data will be made available to anyone outside of study site or not involved in the study.
  However patients will be allocated a study number that will be shared with the participating laboratory and the funder so that data analysis can be done.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: 1 March 2025-15 December 2025
Access Criteria: All data will be kept confidential and at the study site. No IPD will be made available to anyone outside of study site or not involved in the study.
  The laboratory that will be doing the blood sampling analysis and the funder who will be doing the statistics for the study will have access to non-identifiable data for the individual participants
URL: https://www.tamesideandglossopicft.nhs.uk/